CLINICAL TRIAL: NCT01893372
Title: Phase II Study of Eltrombopag With or Without Continuation of Hypomethylating Agent After Hypomethylating Agent Failure For Patients With Myelodysplastic Syndrome (MDS)
Brief Title: Eltrombopag With or Without Hypomethylating Agent After Hypomethylating Agent Failure For Patients With Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: GlaxoSmithKline (Industry); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0225; NCI-2013-02252 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-07-02; First posted 2013-07-09 (Estimated); Results first posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Leukemia
Keywords: Leukemia; Myelodysplastic syndrome; MDS; Overall response rate; ORR; Eltrombopag; Promacta; Hypomethylating Agent
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Eltrombopag (Experimental): Eltrombopag 200 mg by mouth daily in a 28 day cycle.
  Interventions: Drug: Eltrombopag
- Eltrombopag + Hypomethylating Agent (HMA) (Experimental): Eltrombopag in combination with continuation of hypomethylating agent in 28-day cycles. Eltrombopag 200 mg by mouth daily in a 28 day cycle.
  The choice of HMA agent (e.g. azacitidine or decitabine) will be the HMA the patient has received prior to enrollment on study. Eltrombopag should be initiated at the start of the next HMA cycle whenever possible so the start date of both agents is consistent.
  Interventions: Drug: Eltrombopag; Drug: Hypomethylating Agent (HMA)

INTERVENTIONS:
Drug: Eltrombopag — 200 mg by mouth daily in a 28 day cycle.
  Other Names: Promacta
Drug: Hypomethylating Agent (HMA) — The choice of HMA agent (e.g. azacitidine or decitabine) will be the HMA the patient has received prior to enrollment on study.
  Arms: Eltrombopag + Hypomethylating Agent (HMA)

SUMMARY:
The goal of this clinical research study is to learn if eltrombopag can help to control MDS. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to 1 of 2 arms.The selection of treatment arm will be made by you and your treating physician.

* If you are in Arm A, you will receive eltrombopag alone.
* If you are in Arm B, you will receive eltrombopag and will continue to receive the hypomethylating agent that you were receiving before you took part in this study.

Study Drug Administration:

You will take eltrombopag by mouth every day of each 28-day study cycle. If you are in Arm B, you will also continue to take the hypomethylating agent you took before joining the study at the same dosing schedule you were receiving before entering this study.

Eltrombopag should be taken on an empty stomach (1 hour before or 2 hours after a meal). Do not eat calcium-rich foods (such as dairy products and calcium fortified juices), or take other drugs (such as antacids) or supplements containing iron, calcium, aluminum, magnesium, selenium, and/or zinc for 2 hours before or 4 hours after taking eltrombopag. If a dose of eltrombopag is vomited, it should not be made up or re-taken on the same day. If the morning dose is missed, it may be taken up until 5:00 PM on the same day.

Study Visits:

On Day 1 of all Cycles:

* You will have a physical exam including vital signs.
* Blood (about 2-3 teaspoons) will be drawn for routine tests.

On Days 8, 15, and 22 of Cycle 1:

* Your vital signs (blood pressure, heart rate, and temperature) will be measured.
* Blood (about 2-3 teaspoons) will be drawn for routine tests.

If the doctor thinks it is needed, on Day 1 of every 3 cycles (Cycles 3, 6, 9, and so on), you will also have a bone marrow aspirate/biopsy to check the status of the disease and for cytogenetic testing.

Length of Study:

You may continue taking the study drug(s) for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug(s) if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after the follow-up visits.

End-of-Treatment Visit:

Within 5 days of your last dose of study drug, you will come to the clinic for an end-of-treatment visit. The following procedures will be performed:

* You will have a physical exam.
* Blood (about 2-3 teaspoons) will be drawn for routine tests.
* You may have a bone marrow aspirate/biopsy collected to check the status of the disease and for cytogenetic testing.

Follow-up Visit:

About 28 days after your last dose of study drug, you will come to the clinic for a follow-up visit. the following procedures will be performed:

* You will have a physical exam.
* Blood (about 2-3 teaspoons) will be drawn for routine tests.

This is an investigational study. Eltrombopag is FDA approved and commercially available for the treatment of low platelet counts in patients with idiopathic thrombocytopenic purpura (ITP -- a severe bleeding disease). Its use in this study is investigational. Azacitidine and decitabine are each FDA approved for the treatment of MDS and are commercially available. The study doctor can explain how the study drug(s) are designed to work.

Up to 46 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Signed, informed consent must be obtained prior to any study specific procedures.
2. Subjects with a histologically confirmed diagnosis of MDS by FAB criteria, including both MDS and RAEB-T (AML with 20-30% blasts and multilineage dysplasia) by World Health Organization (WHO) classification are eligible.
3. Patients must have completed at least 4 cycles of hypomethylating agent therapy (e.g azacitidine or decitabine) with failure to achieve at least a partial response, or with the presence of ongoing cytopenias per International Working Group (IWG) (platelet count < 100x10^9/L, hemoglobin <11g/L or Absolute Neutrophil Count (ANC) <1x10^9/L). Patients with progressive disease on HMA-therapy prior to this time point are also eligible at the time of documented progression. Therapy with decitabine analogs (i.e. SGI-110) will be considered as decitabine for the purposes of this study.
4. Platelet count <100x10^9/L
5. Low, intermediate-1, intermediate-2 or High-risk category by International Prognostic Scoring System (IPSS)
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
7. Adequate liver function, as evidenced by a serum bilirubin </=2x the ULN (except for patients with a confirmed diagnosis of Gilbert's Disease) and an Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) </=3x the laboratory Upper Limit of Normal (ULN).
8. Serum creatinine </=2x upper limit of normal
9. Subjects must be>/= 18 years of age at the time of informed consent, because no dosing or adverse event data are currently available on the use of eltrombopag in children.
10. Subject is practicing an acceptable method of contraception (documented in chart). Female subjects (or female partners of male subject) must either be of non-childbearing potential (hysterectomy, bilateral oophorectomy, bilateral tubal ligation or post-menopausal > 1 year), or of childbearing potential and use one of the following highly effective methods of contraception (i.e. Pearl index < 1.0%) from 2 weeks prior to administration of study medication, throughout the study, and 28 days after completion or premature discontinuation from the study: - Complete abstinence from intercourse; - Intrauterine device (IUD); - Two forms of barrier contraception (diaphragm plus spermicide, and for males condom plus spermicide); - Male partner is sterile prior to entry into the study and is the only partner of the female; - Systemic contraceptives (combined or progesterone only).
11. Patients must have recovered from acute toxicity (to grade 1 or less) of all previous therapy prior to enrollment. Treatment may start earlier if necessitated by the patient's medical condition (e.g. progressive disease) following discussion with the Investigator.

Exclusion Criteria:

1. Subjects with any prior exposure to a thrombopoietin-receptor agonist
2. Any prior or co-existing medical condition that in the investigator's judgment will substantially increase the risk associated with the subject's participation in the study
3. Psychiatric disorders or altered mental status precluding understanding of the informed consent process and/or completion of the necessary study procedures
4. Active uncontrolled serious infection or sepsis at study enrollment
5. Clinically significant gastrointestinal disorders that may interfere with absorption of drug.
6. History of arterial thrombosis (i.e. stroke) in the past year
7. History of venous thrombosis currently requiring anti-coagulation therapy
8. Unstable angina, congestive heart failure (New York Heart Association (NYHA) > Class II), uncontrolled hypertension (diastolic blood pressure > 100mmHg), or recent (within 1 year) myocardial infarction
9. Subjects with a QTc > 480 msec (QTc > 510 msec for subjects with Bundle Branch Block) at baseline
10. Pregnant or breast-feeding because there are no adequate and well-controlled studies of eltrombopag use in pregnancy and it is unknown whether eltrombopag is excreted in human milk.
11. Subjects with known history of human immunodeficiency virus (HIV) or active infection with hepatitis C virus (HCV) or hepatitis B virus (HBV), because eltrombopag is hepatically cleared, and underlying hepatic impairment may lead to an increased risk of hepatotoxicity. Eltrombopag has not been evaluated with combination antiretroviral regimens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2019-01-06 (Actual); Study Completion 2019-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Courtney DiNardo, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Details: October 2013 to January 2016
Groups:
- Eltrombopag + Hypomethylating Agent (HMA): Eltrombopag in combination with continuation of hypomethylating agent in 28-day cycles. Eltrombopag 200 mg by mouth daily in a 28 day cycle.
  The choice of HMA agent (e.g. azacitidine or decitabine) will be the HMA the patient has received prior to enrollment on study. Eltrombopag should be initiated at the start of the next HMA cycle whenever possible so the start date of both agents is consistent.
  Eltrombopag: 200 mg by mouth daily in a 28 day cycle.
  Hypomethylating Agent (HMA): The choice of HMA agent (e.g. azacitidine or decitabine) will be the HMA the patient has received prior to enrollment on study.
Period: Overall Study
Arm/Group | Eltrombopag | Eltrombopag + Hypomethylating Agent (HMA)
Started | 7 | 22
Completed | 7 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eltrombopag | Eltrombopag + Hypomethylating Agent (HMA) | Total
Number analyzed (Participants) | 7 | 22 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 6
  >=65 years | 5 | 18 | 23
Age, Continuous [Median (Full Range); unit: years] | 74 [61 to 80] | 72 [42 to 84] | 72 [42 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 9 | 12
  Male | 4 | 13 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 6 | 18 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 7 | 22 | 229

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Overall response rate (ORR) based on the International Working Group (IWG)-2006 criteria, which include complete remission (CR), partial remission (PR), and major hematologic improvement (HI). Patients' overall response assessed after at least 2 cycles of treatment and no more than after 6 cycles of treatment and each cycle is 28 days. CR is Bone marrow of </= 5% myeloblasts with normal maturation of cell lines, persistent dysplasia and a hemoglobin >/= 11g/dl, platelets >/= 100x10^9/L, neutrophils >/= 1.0x10^9/L and 0% blasts. PR is the same as CR but bone marrow blasts decreased by >/=50% but still 5% over pre-treatment. HI is described by the number of individually affected cell lines. (E = Erythroid, N = Neutrophils, P = Platelet). HI-E is a 2 gram increase in hemoglobin. HI-N is at least a 100% increase or an absolute increase of more than 500/mm^3. HI-P is an absolute increase of 30/mm^3 or a 50% increase
Time Frame: After second 28 day cycle
Measure: Count of Participants; unit: Participants
Arm/Group | Eltrombopag | Eltrombopag + Hypomethylating Agent (HMA)
Number analyzed (Participants) | 7 | 22
Participants | 0 | 3

2. Primary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) was measured from the time of study enrollment until death from any cause or fate of the last follow-up.
Time Frame: Through study completion. Up to 3 years, 3 months.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Eltrombopag | Eltrombopag + Hypomethylating Agent (HMA)
Number analyzed (Participants) | 7 | 22
Weeks | 57.9 [4.8 to 165.1] | 40.4 [2.3 to 150.4]

3. Secondary Outcome: Number of Participants Transforming From Myelodysplastic Syndrome (MDS) to Acute Myeloid Leukemia (AML)
Time Frame: Up to 3 years, 3 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Eltrombopag | Eltrombopag + Hypomethylating Agent (HMA)
Number analyzed (Participants) | 7 | 22
Participants | 1 | 7

4. Secondary Outcome: Number of Participants Achieving a Platelet Response
Description: Platelet response is Hematologic Improvement with platelet response (HI-P), defined as an absolute increase of >/= 30 x 10^9/L for patients starting with >20 x 10^9/L platelets or increase from <20 x 10^9/L to >20 x 10^9/L and by at least 100%
Time Frame: 3 Years
Measure: Count of Participants; unit: Participants
Arm/Group | Eltrombopag | Eltrombopag + Hypomethylating Agent (HMA)
Number analyzed (Participants) | 7 | 22
Participants | 0 | 3

ADVERSE EVENTS:
Time Frame: Through study completion. Up to 3 years, 3 months.
Arm/Group | Eltrombopag | Eltrombopag + Hypomethylating Agent (HMA)
All-Cause Mortality (participants affected / at risk) | 1/7 | 4/22
Serious Adverse Events (participants affected / at risk) | 3/7 | 16/22
Other Adverse Events (participants affected / at risk) | 1/7 | 16/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eltrombopag (N=7) | Eltrombopag + Hypomethylating Agent (HMA) (N=22)
Abdominal Pain (General disorders) | 1 (1) | 1 (1)
Aenmia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Atrial Fibrillaiton (Cardiac disorders) | 0 (0) | 1 (1)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Death (General disorders) | 0 (0) | 2 (2)
Infection (Infections and infestations) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Febrile Neutropenia (Infections and infestations) | 0 (0) | 4 (5)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lung Infection (Infections and infestations) | 2 (2) | 4 (5)
Neoplasms benigh, malignantand unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Rectal Hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 2 (2)
Device Related Infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eltrombopag (N=7) | Eltrombopag + Hypomethylating Agent (HMA) (N=22)
Fatigue (General disorders) | 1 (1) | 13 (13)
Abcess Under Arm (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Back Pain (General disorders) | 0 (0) | 1 (1)
Bladder Infection (Infections and infestations) | 0 (0) | 1 (1)
Blurred Vision (Eye disorders) | 0 (0) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 7 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Fever (General disorders) | 1 (1) | 3 (5)
Flu Like Symptoms (General disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 1 (1)
Hyperbilirubinemia (Investigations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Intermittent Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intermittent Fatigue (General disorders) | 0 (0) | 1 (1)
Jaundice (Investigations) | 0 (0) | 2 (2)
Joint Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 7 (7)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-23): https://cdn.clinicaltrials.gov/large-docs/72/NCT01893372/Prot_SAP_000.pdf